CLINICAL TRIAL: NCT00836628
Title: A Phase I Study Using Submyeloablative DOsing of Intravenous Busulfan (Busulfex) for Refractory Brain Tumors
Brief Title: Study of Busulfan for Refractory Central Nervous System (CNS) Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Stewart Goldman, Chair of Hem/Onc/Stem Cell, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNS 1100
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Refractory Brain Tumors
MeSH Terms: conditions — Brain Neoplasms | interventions — Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- experimental (Experimental)
  Interventions: Drug: Busulfan

INTERVENTIONS:
Drug: Busulfan
  Other Names: Busulfex ®

SUMMARY:
This protocol is aimed at establishing a maximum tolerated dose (MTD) for submyeloablative doses of Busulfex ® with the hope that a tolerable, submyeloablative dose can be established to test efficacy as alternative therapy for refractory pediatric brain tumors.

DETAILED DESCRIPTION:
Pediatric brain tumors remain among the most common malignancies in childhood, second only to leukemia, representing 20% of all childhood cancers in the United States (1). Although significant strides have been made in therapies for other pediatric malignancies, mortality for patients with brain tumors remains high. The mainstay of therapy for CNS tumors has been a combination of surgery, chemotherapy, and radiation. High dose chemotherapy with stem cell transplant has been proposed as an alternative to radiation, in very young children and for relapsed patients. Stem cell transplantation however is not without significant side effects as well as transplant related mortality.

Busulfan is an alkylating agent and is able to exert its cytotoxic effects through hydrolysis and subsequent production of carbonium ions, directly alkylating DNA, interfering with its replication, and ultimately leading to cell death (2). Busulfan readily crosses the blood barrier, allowing for CNS levels nearly equal to those of plasma levels (5,6).

Primary Objectives:

To determine the maximum tolerated dose (MTD) of Busulfex ® in children with recurrent, progressive, or refractory primary brain tumors.

Secondary Objectives:

To obtain preliminary data regarding progression free survival (PFS) and event free survival (EFS) when Busulfex ® is used at submyeloablative doses in children with recurrent, progressive, or refractory primary brain tumors.

To describe the plasma pharmacokinetics of Busulfex ® in children with recurrent, progressive, or refractory primary brain tumors, using a continuous infusion.

ELIGIBILITY:
Inclusion Criteria:

Age: Age >2 year and ≤ 21 years Histologic Diagnosis Any histological proven (confirmed by institutional pathology report; pathology slides from outside referring outside institutions are not required.) recurrent or progressive CNS tumor. (optic pathway and brainstem gliomas allowed without histologic verification, but must have diagnostic imaging).

Life Expectancy Patients must have a life expectancy of ≥ 2 months. Prior Therapy There is no limit to the number of prior therapies a patient has received

* Must be ≥ 3 weeks from myelosuppressive chemotherapy (6 weeks from nitrosoureas) and have demonstrated recovery (ANC ≥ 1000/uL) from their last course of chemotherapy
* ≥ 6 months following allogeneic stem cell transplantation
* ≥ 3 months following autologous stem cell transplantation
* ≥ 3 months from craniospinal radiation
* ≥ 4 weeks from focal radiation
* ≥ 7 days from any past biologic/immunotherapy
* ≥ 1 week from any hematopoietic growth factors Concomitant Medication
* Patients taking Itraconazole or Phenytoin will be excluded. Patients must be off of these medications for at least 3 days prior to entering this trial. If the patient is taking phenytoin for seizures at the time of study enrollment, it must be stopped at least 3 days prior to starting therapy and Clonazepam will be substituted during the Busulfex ® infusions and for 24 hours following the infusion.
* Patients on growth stimulating factors, such as GCSF, will be allowed to continue these medications only as indicated in the study.
* Patients may be taking steroids while participating in this trial, but should be on a stable dose for >1 week prior to enrollment.
* Medications interacting with the CYP3A4 substrate should also be avoided while the patient is on study.
* Patients should also be on Pneumocystis prophylaxis while participating in this study. Pentamidine will be required, with a recommended dose of 4 mg/kg given intravenously every month. Pentamidine should continue throughout the duration of the trial.

Organ Function Requirements Adequate Bone Marrow Function Defined As

* Peripheral absolute neutrophil count (ANC) greater than or equal to 1000/ul (off growth factors x 48 hrs)
* Platelet count greater than or equal to 100,000/uL (transfusion independent)
* Hemoglobin greater than or equal to 8.0 gm/dL (may receive RBC transfusions) Adequate Renal Function Defined As
* Serum creatinine less than or equal to 1.5 x upper limit of normal, or
* Estimated creatinine clearance GFR greater than or equal to 70 ml/min/1.73 m² by the Schwartz formula Adequate Liver Function Defined As
* Total bilirubin within normal range
* SGPT (ALT) within normal range Adequate Pulmonary Function Defined As
* Oxygen saturation >92% on room air Central Nervous System Function Defined As
* Patients with seizure disorder may be enrolled; Patients MUST be on an anti-seizure medication upon enrollment, but this medication CANNOT be phenytoin or carbamezepine.
* Patients must not be in status, coma or assisted ventilation prior to study enrollment.
* Stable neurologic exam of at least 1 week duration Performance Level Karnofsky/ Lansky 50 or greater

Exclusion Criteria:

* Pregnancy/Contraception: patients who are pregnant or breast-feeding will not be eligible.
* Patients of childbearing potential must practice an effective method of birth control while participating on the study.
* Females > 13 years of age or those who have achieved menarche must have a negative pregnancy test prior to study entry.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Goldman, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago

IPD SHARING:
Plan to Share IPD: Undecided